CLINICAL TRIAL: NCT00665899
Title: A Couples Approach to Enhance Breast Cancer Survivorship
Acronym: CanThrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 04-0977; 1R01CA107477-01 (NIH); LCC 0402 (Other: UNC)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Early-Stage Breast Cancer
Keywords: breast cancer; couples; cognitive behavioral therapy; Women with early stage breast cancer and their partners.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cancer-Focused Relationship Enhancement (Experimental): Cancer-Focused Relationship Enhancement
  Interventions: Behavioral: Cancer-Focused Relationship Enhancement
- Couple's Cancer Education (Experimental): Couple's Cancer Education
  Interventions: Behavioral: Couple's Cancer Education
- Usual Care (No Intervention): Cancer-Related Community and Internet Resources

INTERVENTIONS:
Behavioral: Cancer-Focused Relationship Enhancement — Couples meet individually with a health educator for 6 sessions to learn about ways to support each other and communicate about breast cancer related issues.
  Arms: Cancer-Focused Relationship Enhancement
Behavioral: Couple's Cancer Education — Couples meet individually with a health educator for 6 sessions to discuss the medical aspects of breast cancer and treatment options.
  Arms: Couple's Cancer Education

SUMMARY:
The purpose of the proposed study is to evaluate the efficacy of a new couple-based intervention for women with recently diagnosed, early stage breast cancer and their spouses or male partners. This cancer-focused relationship enhancement intervention adapts well-validated cognitive-behavioral interventions to teach patients and partners specific relationship skills, such as problem-solving skills, communication, and maximizing positive interactions, that they can use in addressing breast cancer. This project's major goals are to improve the patient's individual functioning and specific aspects of the couple's relationship affected by breast cancer (e.g., mood, role functioning, sexual functioning, and social support). In the current investigation, cancer-focused relationship enhancement will be compared to (a) a couple-based Cancer Education intervention and (b) a Treatment-as-Usual condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early stage breast cancer within last year
* No history of breast cancer, or other cancers in last 5 years (except skin cancer)
* Living together in a committed heterosexual relationship
* read and speak English
* Agree to participate

Exclusion Criteria:

* Stage 3b and above breast cancer
* Notable psychopathology, including severe depression with suicidality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2004-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Relationship Functioning, Individual Functioning, Cancer Related Physical Functioning | Pre, post, 6 month follow-up, 12 month follow-up

SECONDARY OUTCOMES:
Observational coding of couples social support and decision making conversations | pre, post, 6 month follow-up, 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Baucom, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill; Laura S Porter, Ph.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Zimmermann T, Heinrichs N, Baucom DH. "Does one size fit all?" moderators in psychosocial interventions for breast cancer patients: a meta-analysis. Ann Behav Med. 2007 Nov-Dec;34(3):225-39. doi: 10.1007/BF02874548. PMID 18020933
- [Background] Baucom DH, Porter LS, Kirby JS, Gremore TM, Keefe FJ. Psychosocial issues confronting young women with breast cancer. Breast Dis. 2005-2006;23:103-13. doi: 10.3233/bd-2006-23114. PMID 16823173
- See also: CanThrive Website — http://www.canthrive.org